CLINICAL TRIAL: NCT02995629
Title: Patient Comfort Using Green (532 nm) Versus Yellow (577 nm) Laser Indirect Ophthalmoscopy Panretinal Photocoagulation for Proliferative Diabetic Retinopathy
Brief Title: Patient Comfort Using Green vs. Yellow Pan Retinal Photocoagulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wills Eye (Other)
Collaborators: Mid Atlantic Retina (Other)
Responsible Party: Principal Investigator, MidAtlantic Retina, Dr. Allen Chiang, MD, Wills Eye
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 16-560
Record Dates: First submitted 2016-12-05; First posted 2016-12-16 (Estimated); Last update posted 2016-12-16 (Estimated); Status verified 2016-12

CONDITIONS: Proliferative Diabetic Retinopathy - High Risk

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- green (532 nm) laser (Experimental): scatter laser indirect ophthalmoscopy pan retinal photocoagulation
  Interventions: Procedure: laser indirect ophthalmoscopy pan retinal photocoagulation
- yellow (577 nm) laser (Experimental): scatter laser indirect ophthalmoscopy pan retinal photocoagulation
  Interventions: Procedure: laser indirect ophthalmoscopy pan retinal photocoagulation

INTERVENTIONS:
Procedure: laser indirect ophthalmoscopy pan retinal photocoagulation — * Prior to procedure, eligible patient is dilated and a topical anesthesia is administered 3 to 5 minutes prior to treatment initiation
  * Treatment duration is fixed at 50 minutes and power is titrated until moderate gray-white burns are achieved, avoiding long ciliary nerves
  * Target treatment of 250 spots
  * Only one eye per eligible patient randomized with regard to whether green or yellow laser utilized first
  * After treatment,pain assessment conducted:spot count, laser parameters and treatment duration recorded for each respective laser wavelength
  Other Names: PRP laser

SUMMARY:
Our aim is to compare patient comfort when using the 532 nanometer (green) wavelength laser to the 577 nanometer (yellow) wavelength laser during pan retinal photocoagulation to treat patients with diabetic retinopathy. Secondary outcome measures will be power (mW) required to achieve gray-white retinal burns and duration of treatment.

DETAILED DESCRIPTION:
As demonstrated in the Diabetic Retinopathy Study (DRS), panretinal photocoagulation (PRP) reduces the risk of severe vision loss in patients with proliferative diabetic retinopathy. The DRS recommended that PRP treatment consist of 1,200 - 1,600 laser burns 500 µm in size, one half to one burn width apart, applied to the peripheral retina in a scatter fashion. Most patients who undergo PRP experience discomfort/pain during the procedure. Once present, pain can affect the number and quality of burns delivered and can indirectly increase the number of sessions required to complete the therapy.This may in turn adversely affect patient compliance. Although retrobulbar and peribulbar blocks can provide adequate anesthesia for PRP, these anesthetic methods carry rare but serious risks such as retrobulbar hemorrhage. Previous studies have explored other ways to reduce discomfort related to PRP, including optimization of laser settings, oral and topical analgesics, subconjunctival anesthesia, and even acupuncture.

Currently, green lasers (521 - 532 nm wavelength) are most commonly utilized for performing PRP in clinical practice. Yellow lasers (577 nm wavelength) have been of recent interest in treating diabetic macular edema with micropulse subthreshold grid photocoagulation, but have not been extensively studied in PRP for diabetic retinopathy. Compared to shorter wavelength laser, yellow laser comports high transmission through dense ocular media and less light scattering than shorter wavelengths which minimizes spot size and reduces thermal spread. The limited literature comparing green and yellow laser for PRP in diabetic retinopathy has shown that yellow laser requires less power to achieve a retinal burn. In theory this should translate into a reduction in perceived pain experienced during PRP, however a comparison of green and yellow lasers in this regard has not yet been directly examined and quantified.

ELIGIBILITY:
Inclusion Criteria:

* patient of Wills Eye Hospital Retina Service and/or Mid Atlantic Retina
* volunteer patients age 18 years and older.
* healthy enough to participate in the study.
* willing and able to consent to participation in the study.
* diagnosis of PDR with HRC based on clinical criteria outlined by the DRS.

Exclusion Criteria:

* patient less than 18 years of age
* institutionalized patient
* prisoner
* significant media opacity obscuring a view of the superior retina
* history of intra-ocular surgery except cataract surgery
* history of PRP laser within the last 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-03; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Perceived patient pain assessment | a single time point within 2 minutes of completing laser treatment
  Assessed using a standardized Wong-Baker faces pain scale

SECONDARY OUTCOMES:
Minimum power requirement to achieve moderate gray-white retinal burns | During treatment
Time of treatment | During treatment
  Time required to treat with each laser

CONTACTS AND LOCATIONS:
Overall Officials: Allen Chiang, MD, Principal Investigator — Mid Atlantic Retina
Locations (1):
- Mid Atlantic Retina- Wills Eye Institute, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Manuscript is under development.

REFERENCES:
- [Background] Photocoagulation treatment of proliferative diabetic retinopathy. Clinical application of Diabetic Retinopathy Study (DRS) findings, DRS Report Number 8. The Diabetic Retinopathy Study Research Group. Ophthalmology. 1981 Jul;88(7):583-600. PMID 7196564
- [Background] Richardson C, Waterman H. Pain relief during panretinal photocoagulation for diabetic retinopathy: a national survey. Eye (Lond). 2009 Dec;23(12):2233-7. doi: 10.1038/eye.2008.421. PMID 19169228
- [Background] Alvarez-Verduzco O, Garcia-Aguirre G, Lopez-Ramos Mde L, Vera-Rodriguez S, Guerrero-Naranjo JL, Morales-Canton V. Reduction of fluence to decrease pain during panretinal photocoagulation in diabetic patients. Ophthalmic Surg Lasers Imaging. 2010 Jul-Aug;41(4):432-6. doi: 10.3928/15428877-20100525-02. Epub 2010 May 28. PMID 20608612
- [Background] Mirshahi A, Lashay A, Roozbahani M, Fard MA, Molaie S, Mireshghi M, Zaferani MM. Pain score of patients undergoing single spot, short pulse laser versus conventional laser for diabetic retinopathy. Graefes Arch Clin Exp Ophthalmol. 2013 Apr;251(4):1103-7. doi: 10.1007/s00417-012-2167-5. Epub 2012 Oct 11. PMID 23052718
- [Background] Wu WC, Hsu KH, Chen TL, Hwang YS, Lin KK, Li LM, Shih CP, Lai CC. Interventions for relieving pain associated with panretinal photocoagulation: a prospective randomized trial. Eye (Lond). 2006 Jun;20(6):712-9. doi: 10.1038/sj.eye.6701989. Epub 2005 Jul 8. PMID 16021194
- [Background] Ko BW, Shim JH, Lee BR, Cho HY. Analgesic effects of tramadol during panretinal photocoagulation. Korean J Ophthalmol. 2009 Dec;23(4):273-6. doi: 10.3341/kjo.2009.23.4.273. Epub 2009 Dec 4. PMID 20046687
- [Background] Zakrzewski PA, O'Donnell HL, Lam WC. Oral versus topical diclofenac for pain prevention during panretinal photocoagulation. Ophthalmology. 2009 Jun;116(6):1168-74. doi: 10.1016/j.ophtha.2009.01.022. Epub 2009 Apr 19. PMID 19376588
- [Background] Tesha PE, Giavedoni LR, Berger AR, Altomare F, Chow DR, Navajas EV, Yoganathan P, Wong DT, Principe A. Subconjunctival lidocaine before laser treatment: a randomized trial. Ophthalmology. 2010 Sep;117(9):1810-4. doi: 10.1016/j.ophtha.2010.01.036. Epub 2010 Jun 8. PMID 20570360
- [Background] Chiu HH, Wu PC. Manual acupuncture for relieving pain associated with panretinal photocoagulation. J Altern Complement Med. 2011 Oct;17(10):915-21. doi: 10.1089/acm.2010.0082. Epub 2011 Oct 6. PMID 21978192
- [Background] Vujosevic S, Martini F, Longhin E, Convento E, Cavarzeran F, Midena E. SUBTHRESHOLD MICROPULSE YELLOW LASER VERSUS SUBTHRESHOLD MICROPULSE INFRARED LASER IN CENTER-INVOLVING DIABETIC MACULAR EDEMA: Morphologic and Functional Safety. Retina. 2015 Aug;35(8):1594-603. doi: 10.1097/IAE.0000000000000521. PMID 25719988
- [Background] Yadav NK, Jayadev C, Mohan A, Vijayan P, Battu R, Dabir S, Shetty B, Shetty R; Medscape. Subthreshold micropulse yellow laser (577 nm) in chronic central serous chorioretinopathy: safety profile and treatment outcome. Eye (Lond). 2015 Feb;29(2):258-64; quiz 265. doi: 10.1038/eye.2014.315. Epub 2015 Jan 23. PMID 25613846
- [Background] Mainster MA. Wavelength selection in macular photocoagulation. Tissue optics, thermal effects, and laser systems. Ophthalmology. 1986 Jul;93(7):952-8. doi: 10.1016/s0161-6420(86)33637-6. PMID 3763141